CLINICAL TRIAL: NCT01499550
Title: Nocturnal Transnasal Insufflation in Patients With COPD and Hypercapnia
Brief Title: Nocturnal Transnasal Insufflation (nTNI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: TNI Medical AG (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Head of the Department of pneumology at Helios Klinik Ambrock, Institut für Pneumologie Hagen Ambrock eV
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: nTNI2011
Record Dates: First submitted 2011-11-03; First posted 2011-12-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: COPD; Hypercapnia
Keywords: transnasal high flow therapy; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNI application (Experimental): In this study arm the patient is treated with humidified transnasal high flow (TNI) plus oxygen (result flow: 20 L/min).
  Interventions: Device: humidified transnasal insufflation (TNI20oxy)
- Oxygen treatment (Active Comparator): Long term oxygen treatment (LOT) is the routine treatment in patients suffering from COPD. In this study arm the patient is treated with his individual oxygen flow rate.
  Interventions: Other: overnight oxygen treatment with individual flow rate

INTERVENTIONS:
Device: humidified transnasal insufflation (TNI20oxy) — The alternative breathing support with TNI supplies COPD patients with 20L/min of warm humidified air. This method may be applicable to wash out the dead space between glottis and nasal opening. Pre-investigations have shown that 45 minutes of TNI during daytime reduced PCO2 and respiratory rate compared to application of oxygen alone.Transcutaneous PCO2 is measured over night. A capillary blood gas analysis (BGA) is carried out at beginning and end of each measurement night.
  Other Names: TNI20oxy
  Arms: TNI application
Other: overnight oxygen treatment with individual flow rate — The patient is treated with his individual oxygene flow rate. Transcutaneous PCO2 is measured over night. A capillary blood gas analysis (BGA) is carried out at beginning and end of each measurement night.
  Arms: Oxygen treatment

SUMMARY:
On the basis of different studies the long term oxygen treatment is deemed to be routine treatment in patients suffering from chronic obstructive pulmonary disease (COPD) at appearance of hypoxaemia. Non invasive ventilation (NIV) is the treatment of choice in hypercapnic COPD patients with respiratory acidosis at acute respiratory decompensation. Several prospective randomized studies have shown a reduction of acute mortality as result. But everyday practice shows that COPD patients with chronic hypercapnia hardly accustom oneself to nocturnal ventilation. Reasons are not known yet, but substantial pulmonary overinflation or the appearance of depressions or rather anxiety disorders are possible causes. On the other hand patients may not notice any subjective improvement of symptoms and won't accept the burden of a tight fitting mask during the night. The aim of the present study is to determine the effect on gas exchange of a nocturnal transnasal application of an oxygen-enriched gaseous mixture via nasal cannula and the subjective acceptance. This is compared to a nocturnal transnasal application of oxygen alone in randomized order for at least 6 hours each night.

Thirty hypercapnic COPD GOLD IV patients (PCO2 > 50 mmHg) will be included. The two night Polysomnographies (PSG) will be evaluated with special attention to nasal flow measurements, breathing effort, oxygen saturation and an additional transcutaneous PCO2 measurement. At begin and end of each measurement night a capillary blood gas analysis is made.

ELIGIBILITY:
Inclusion Criteria:

* Hypercapnia in Routine Blood Gas Analysis with > 50 mmHg PCO2
* Clinically stable respiratory situation
* Treatment on normal ward possible

Exclusion Criteria:

* Before known obstructive sleep apnea syndrome (OSA)
* A found OSA during study means no exclusion
* Any other severe or acute physical illness which requires intensive medical care
* Acute hypercapnic decompensation with pH < 7.30 in capillary Blood Gas Analysis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
PCO2 decrease | within 2 days
  During the study nights the patients PCO2 value is measured transcutaneous as well as by capillary blood gas analyses (BGA) in the evening and in the morning. The differences in PCO2 values of the morning BGA will be compared, a PCO2 decrease is supposed to be assessed under TNI treatment.

SECONDARY OUTCOMES:
Changes of breathing pattern | within 2 days
  Changes of breathing pattern and breahing frequency will be recorded during the nights and means and course evaluated. Breathing Frequency is supposed to decrease under TNI treatment

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen Ambrock, Ambrocker Weg 60, D58091 Hagen
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany